CLINICAL TRIAL: NCT01106209
Title: Neutrophil Extracellular Trap Formation in Newborn Infants at Risk for Inflammatory Syndromes
Status: Terminated | Type: Observational
Why Stopped: Lack of enrollment
Sponsor: University of Utah (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: 119244; R01HD093826 (NIH)
Record Dates: First submitted 2010-04-15; First posted 2010-04-19 (Estimated); Results first posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2022-11

CONDITIONS: Prematurity; Necrotizing Enterocolitis
Keywords: premature infants; polymorphonuclear leukocytes; PMNs; neutrophil extracellular traps; NET formation; necrotizing enterocolitis
MeSH Terms: conditions — Premature Birth; Enterocolitis, Necrotizing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and intestinal tissue samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Prematurely born infants in the NICU: Preterm infant patients delivered at UUMC and hospitalized in the NICU who are ≤1500 grams or <30 weeks gestational age at birth.
- Healthy term infants: Term infants delivered at UUMC without complication, either via cesarean section or vaginal delivery
- Subset: Enrolled preterm infants having surgery at <1 year old for NEC: Enrolled preterm infants who require surgery for NEC within their first year of life for

SUMMARY:
The purpose of this study is to characterize the time to maturation of neutrophil extracellular trap(NET) formation capability in polymorphonuclear leukocytes(PMNs) isolated from newborn premature and term infants. Preterm infants who are enrolled into the study who then go on to require surgery <1 year due to surgical NEC, will have the NET formation reassessed. This study will also determine whether NETs contribute to the pathogenesis of necrotizing enterocolitis (NEC). We hypothesize that NET formation contributes to the pathogenesis of NEC by inappropriately releasing degradative proteins and tissue destructive enzymes into the inflammatory milieu of the premature infant gastrointestinal tract following bacterial translocation. We also hypothesize that the delay in NEC development in premature infants (3rd - 4th week of life) as compared to at-risk term infants (1st week of life) results from a developmental delay in PMN ability to form NETs.

DETAILED DESCRIPTION:
Prematurely born infants are at risk for necrotizing enterocolitis (NEC), the most common gastrointestinal emergency encountered in the newborn intensive care unit. This disease occurs in between 5 - 10% of infants born at less than 30 weeks gestation or less than 1500 grams birth weight. In these patients, NEC routinely develops during the 3rd or 4th week of life. NEC rarely occurs in infants born closer to term; for these patients NEC usually develops during the 1st week of life. So far, no one has explained the inverse relationship between gestational age at birth and the delay in NEC development.

Recently, our laboratory described for the first time an inherent deficiency of innate immunity in newborn infants - failure of neutrophil extracellular trap formation. Neutrophil extracellular traps or NETs are complex lattices of extracellular chromatin and DNA decorated with anti-microbial proteins and degradative enzymes which trap and kill microbes. When the neutrophils of newborn infants develop the ability to form NETs and whether the maturation of NET formation correlates with development of NEC in at risk infants remains unknown.

We have therefore undertaken the following study best described as a prospective, in vitro longitudinal cellular biology study of LPS/PAF-stimulated PMNs isolated from the cord and peripheral blood of premature infants at risk for NEC and from term infants not considered at risk for NEC. We will also assay for NET formation in gastrointestinal tissue samples obtained at the time of surgery for severe NEC in enrolled prematurely born infants. These studies are the first of their kind and aim to answer these important questions.

ELIGIBILITY:
Inclusion Criteria:

1. Preterm infant patients delivered at UUMC and hospitalized in the NICU who are ≤ 1500 grams or <30 weeks gestational age at birth
2. Term infants delivered at UUMC without complication, either via cesarean section or vaginal delivery

Exclusion Criteria:

* No other exclusion criteria

Max Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Preterm and healthy term infants born at the University of Utah Hospital. A subset of preterm infants needing surgery <1 year of age, will be reassessed.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2010-04 (Actual); Primary Completion 2020-06-22 (Actual); Study Completion 2020-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christian C Yost, MD, Principal Investigator — University of Utah
Locations (2):
- United States (2):
  - University of Utah, Salt Lake City, Utah
  - Primary Children's Medical Center, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No infants required surgery during the first year of life, therefore no participants were evaluated in the surgical cohort
Groups:
- Infants Having Surgery at <1 Year Old: Infants who require surgery within their first year of life for NEC
Period: Overall Study
Arm/Group | Prematurely Born Infants in the NICU | Healthy Term Infants | Infants Having Surgery at <1 Year Old
Started | 11 | 3 | 0
Completed | 11 | 3 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: None of our recruited prematurely born infants in the NICU required surgery in the first year of life.
Groups:
- Subset: Enrolled Preterm Infants Having Surgery at <1 Year Old: Enrolled preterm infants who require surgery within their first year of life
- Total: Total of all reporting groups
Arm/Group | Prematurely Born Infants in the NICU | Healthy Term Infants | Subset: Enrolled Preterm Infants Having Surgery at <1 Year Old | Total
Number analyzed (Participants) | 11 | 3 | 0 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11 | 3 | 0 | 14
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: Day] | 1 [1 to 1] | 1 [1 to 1] |  | 1 [1 to 1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 1 |  | 7
  Male | 5 | 2 |  | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 |  | 2
  Not Hispanic or Latino | 9 | 3 |  | 12
  Unknown or Not Reported | 0 | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 |  | 0
  Asian | 0 | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 |  | 0
  Black or African American | 0 | 0 |  | 0
  White | 11 | 3 |  | 14
  More than one race | 0 | 0 |  | 0
  Unknown or Not Reported | 0 | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 3 |  | 14

OUTCOME MEASURES:

1. Primary Outcome: Time to Maturation of Neutrophil Extracellular Trap(NET) Formation
Description: The objective is to characterize the time to maturation of NET formation capability in polymorphonuclear leukocytes(PMNs)isolated from newborn infants.
Time Frame: 60 days
Population: No study participants required surgery during the first year of life.
Measure: Mean (Full Range); unit: Days
Groups:
- Infants Having Surgery at <1 Year Old: Infants admitted to the PCMC same-day surgery unit in preparation for elective surgery within the first year of life
Arm/Group | Prematurely Born Infants in the NICU | Healthy Term Infants | Infants Having Surgery at <1 Year Old
Number analyzed (Participants) | 11 | 3 | 0
Days | 14 [3 to 17] | 5 [4 to 14] |

ADVERSE EVENTS:
Time Frame: First 2 months of life.
Description: Not a clinical study. NEC was a complication of prematurity, not a complication of our observational study.
Groups:
- Infants Having Surgery at <1 Year Old: Infants who go on to have surgery at <1 year of age will have NET formation reassessed. No enrolled infants required surgery at < 1 year of age
Arm/Group | Prematurely Born Infants in the NICU | Healthy Term Infants | Infants Having Surgery at <1 Year Old
All-Cause Mortality (participants affected / at risk) | 1/11 | 0/3 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/3 | 0/0
Other Adverse Events (participants affected / at risk) | 0/11 | 0/3 | 0/0

LIMITATIONS AND CAVEATS:
This is an observational study designed to evaluate NEC incidence with in vitro assessment of neutrophil neutrophil extracellular trap formation. There are too few study participants to draw any meaningful correlations between in vitro NET formation by participant neutrophils and the incidence of NEC in this at-risk population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-15): https://cdn.clinicaltrials.gov/large-docs/09/NCT01106209/Prot_SAP_000.pdf